CLINICAL TRIAL: NCT02427737
Title: Amelioration of Claustrophobia and Disruptive Patient Motion in MRI Imaging (Phase 2 Randomized Training of Sites)
Brief Title: Comfort Talk and Economic Outcomes in MRI
Acronym: ComfortTalk®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hypnalgesics, LLC (Industry)
Collaborators: Ohio State University (Other); Duke University (Other)
Responsible Party: Principal Investigator, Elvira V. Lang, MD, CEO, Hypnalgesics, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2CTOSUD2015
Record Dates: First submitted 2015-04-20; First posted 2015-04-28 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Claustrophobia; Complication of Diagnostic Procedure
Keywords: Magnetic Resonance Imaging; Patient satisfaction; Diagnostic Imaging
MeSH Terms: conditions — Claustrophobia; Patient Satisfaction | interventions — Dosage Forms

STUDY DESIGN:
Intervention Model Description: The original model was to have parallel randomized MRI sites. This was possible at one participating institution, The Ohio State Universty Medical Center (OSU). For the second institution (Duke University) staff cuts resulted in personnel cross-over between test and control sites making randomization impossible. Therefore a sequential model was used compared data from the pre- to post training period for the Duke sites. In total 12 MRI entities contributed, six at OSU, and six at Duke. Also, Duke and OSU turned out to have different modes of data collection. OSU had fully automated capture of patients scheduled, showing, and completing their examination as well as a priori numbers of available imaging slots per time unit. Duke did not collect these data electronically so that personnel could only gather the pertinent measures by daily manual diary entry. Thus the mode of result presentation is not concordant in some aspects among sites.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Comfort Talk® Training (Experimental): In the experimental group, MRI personnel is trained to use Comfort Talk® to help patients who are claustrophobic, anxious, and/or cannot lie still to complete their tests at the onset of the MRI scan.
  Interventions: Behavioral: Comfort Talk® Training
- Control (No Intervention): MRI sites not trained in Comfort Talk®.

INTERVENTIONS:
Behavioral: Comfort Talk® Training — Personnel of MRI units is trained in advanced rapport skills, patient-centered and hypnoidal language, correct use of suggestions and skills of tension diffusion. This entails 16 hrs classroom work, additional on-site post-training support, and access to a post-training support web module resulting in at least 20 hrs training.
  Other Names: Self-hypnotic relaxation; Nonpharmacologic analgesia; Nonpharmacologic anxiolysis; Patient sedation without medication
  Arms: Comfort Talk® Training

SUMMARY:
Annually, an estimated 700,000 patients do not complete their scheduled MRI scans because of claustrophobia or inability to hold still. Training staffs working in MRI facilities to provide Comfort Talk® will enable patients to complete high quality imaging without medication, which will increase satisfaction and comfort while reducing sedation risks for patients, and increase efficiency and reduce loss of revenue for facilities. The effect of such training will be tested at 12 MRI sites in a randomized design. Outcome data will be collected for one year.

DETAILED DESCRIPTION:
Claustrophobia and disruptive patient motion are common impediments to MRI examination, but they may be prevented or ameliorated with a non-pharmacologic behavioral intervention administered by trained staff. The potential benefits of such an intervention are highly significant, considering that the alternatives are to cancel the study or administer sedation. Inability to complete their MRI scans adversely affects an estimated 700,000 patients every year in the US. These patients are either deprived of a diagnosis, subject to diagnostic delays and interpretation errors due to motion artifact, or are exposed to risks of pharmacologic sedation, including death. The imaging facilities typically cannot fill the suddenly vacated examination slots in time before the next scheduled patient and incur considerable lost revenue and efficiency. A negative patient experience further jeopardizes Value-Based reimbursement by the Centers for Medicare and Medicaid Services (CMS) towards which patient satisfaction counts 30%. The long term goal is to provide a validated, clinically feasible means for non-pharmacologic amelioration of claustrophobia and disruptive patient motion, achieved by training facility staff in Comfort Talk®.

Comfort Talk® training consists of a proprietary, standardized R3 Process of Rapport, Relaxation, and Reframing including 2 x 8-hrs class-room interaction, onsite coaching, and institution-specific web-based support to help the MRI team to further develop its own language style and skill set.

The effect of Comfort Talk® training will be quantified in a prospective randomized design at 12 MRI satellites of the Ohio State University Medical Center and Duke University Medical Center. Return of investment of training will be based on a decision-analysis model with focus on number of scans performed, cancellations from no-shows and refusals; patients unable to start or complete a scan; and sedation rates in relation to capacity, cost, and reimbursement schedule. Patient satisfaction scores will be compared using Press Ganey national benchmark percentile rankings and CMS quality standards.

ELIGIBILITY:
Inclusion Criteria:

* Must routinely perform MRI examinations
* Must capture data on noncompletion of MRI scans

Exclusion Criteria:

* No dedicated MRI unit
* Unable to reliably capture data on noncompletion of MRI scans

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elvira V Lang, MD, Principal Investigator — Hypnalgesics, LLC
Locations (3):
- United States (3):
  - Hypnalgesics, LLC, Brookline, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lang EV, Ward C, Laser E. Effect of team training on patients' ability to complete MRI examinations. Acad Radiol. 2010 Jan;17(1):18-23. doi: 10.1016/j.acra.2009.07.002. Epub 2009 Sep 5. PMID 19734060
- [Background] Lang EV, Yuh WT, Ajam A, Kelly R, Macadam L, Potts R, Mayr NA. Understanding patient satisfaction ratings for radiology services. AJR Am J Roentgenol. 2013 Dec;201(6):1190-5; quiz 1196. doi: 10.2214/AJR.13.11281. PMID 24261356
- [Background] Lang EV. A Better Patient Experience Through Better Communication. J Radiol Nurs. 2012 Dec 1;31(4):114-119. doi: 10.1016/j.jradnu.2012.08.001. PMID 23471099
- [Background] Flory N, Lang EV. Distress in the radiology waiting room. Radiology. 2011 Jul;260(1):166-73. doi: 10.1148/radiol.11102211. Epub 2011 Apr 7. PMID 21474702
- [Background] Lang EV, Hatsiopoulou O, Koch T, Berbaum K, Lutgendorf S, Kettenmann E, Logan H, Kaptchuk TJ. Can words hurt? Patient-provider interactions during invasive procedures. Pain. 2005 Mar;114(1-2):303-9. doi: 10.1016/j.pain.2004.12.028. Epub 2005 Jan 26. PMID 15733657
- [Background] Lang EV, Rosen MP. Cost analysis of adjunct hypnosis with sedation during outpatient interventional radiologic procedures. Radiology. 2002 Feb;222(2):375-82. doi: 10.1148/radiol.2222010528. PMID 11818602
- [Background] Lang EV, Benotsch EG, Fick LJ, Lutgendorf S, Berbaum ML, Berbaum KS, Logan H, Spiegel D. Adjunctive non-pharmacological analgesia for invasive medical procedures: a randomised trial. Lancet. 2000 Apr 29;355(9214):1486-90. doi: 10.1016/S0140-6736(00)02162-0. PMID 10801169
- [Background] Norbash A, Yucel K, Yuh W, Doros G, Ajam A, Lang E, Pauker S, Mayr N. Effect of team training on improving MRI study completion rates and no-show rates. J Magn Reson Imaging. 2016 Oct;44(4):1040-7. doi: 10.1002/jmri.25219. Epub 2016 Apr 6. PMID 27126735
- [Result] Ajam AA, Nguyen XV, Kelly RA, Ladapo JA, Lang EV. Effects of Interpersonal Skills Training on MRI Operations in a Saturated Market: A Randomized Trial. J Am Coll Radiol. 2017 Jul;14(7):963-970. doi: 10.1016/j.jacr.2017.03.015. Epub 2017 Apr 28. PMID 28461168
- [Result] Ladapo JA, Spritzer CE, Nguyen XV, Pool J, Lang E. Economics of MRI Operations After Implementation of Interpersonal Skills Training. J Am Coll Radiol. 2018 Dec;15(12):1775-1783. doi: 10.1016/j.jacr.2018.01.017. Epub 2018 Mar 9. PMID 29530323

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At OSUMC randomization was maintained (3 trained, 3 control sites). At Duke University considerable staff cuts at the onset of the trial resulted in extensive staff rotations making maintenance of randomization impossible. Thus a pre-post training comparison for the 6 sites was done (pre-training baseline = control, post-training = training arm)
Pre-assignment Details: Different participants were assessed at baseline and at each period after training.
  Clinical sites, not participants, were enrolled in the study. Note that "participants" refers to all patients scheduled to be examined on the available imaging slots, including patients who showed ("completed") and those who were no-shows ("not completed").
Units Other Than Participants: Imaging slots
Groups:
- Comfort Talk® Training: MRI clinical sites form the experimental group. Their personnel is trained to use Comfort Talk® to help patients who are claustrophobic, anxious, and/or cannot lie still to complete their tests at the onset of the study.
  Comfort Talk® Training: Personnel of MRI units is trained in advanced rapport skills, patient-centered and hypnoidal language, correct use of suggestions and skills of tension diffusion. This will entail 16 hrs classroom work, additional on-site post-training support, and access to a post-training support web module resulting in at least 20 hrs training.
- Control: MRI sites are not be trained in Comfort Talk®.
  Please note that at OSU both trained and control sites had a baseline and three post-training periods.
  At Duke, the data in the initial baseline period became the control data in a pre to post comparison for reasons explained above. Therefore Duke has only 2 time periods with the initial "Baseline" entered as "Control."
Period: OSU Baseline Q4FY15
Arm/Group | Comfort Talk® Training | Control
Started | 4158; 4754 Imaging slots | 3446; 4219 Imaging slots
Completed | 3940; 4754 Imaging slots | 3230; 4219 Imaging slots
Not Completed | 218; 0 Imaging slots | 216; 0 Imaging slots
Period: OSU Q1FY16 (First Post-Training Quarter)
Arm/Group | Comfort Talk® Training | Control
Started | 4030; 4583 Imaging slots | 3246; 4144 Imaging slots
Completed | 3815; 4583 Imaging slots | 3032; 4144 Imaging slots
Not Completed | 215; 0 Imaging slots | 214; 0 Imaging slots
Period: OSU Q2FY16(Second Post Training Quarter)
Arm/Group | Comfort Talk® Training | Control
Started | 4121; 4659 Imaging slots | 3070; 4204 Imaging slots
Completed | 3907; 4659 Imaging slots | 2857; 4204 Imaging slots
Not Completed | 214; 0 Imaging slots | 213; 0 Imaging slots
Period: OSU Q3FY16 (Third Post Training Quarter)
Arm/Group | Comfort Talk® Training | Control
Started | 4148; 4647 Imaging slots | 2931; 4199 Imaging slots
Completed | 3928; 4647 Imaging slots | 2716; 4199 Imaging slots
Not Completed | 220; 0 Imaging slots | 215; 0 Imaging slots
Period: Duke Pre- and Post-Training Groups
Arm/Group | Comfort Talk® Training | Control
Started | 9658; 9658 Imaging slots (Note this is a pre-training to post-training comparison.) | 4446; 4446 Imaging slots (Note Control=Baseline)
Completed | 8879; 9658 Imaging slots | 4051; 4446 Imaging slots
Not Completed | 779; 0 Imaging slots | 395; 0 Imaging slots

BASELINE CHARACTERISTICS:
Population: We obtained cumulative data on equipment utilization represented by the number of patients (participants) examined on a given number of imaging slots available at the MRI units in the time period assessed. Thus no individual data on age, gender, ethnicity are available, reducing the population analyzable for these characteristics to zero.
Units Other Than Participants: Imaging Slots
Groups:
- Comfort Talk® Training OSU: Three MRI clinical sites form the experimental group at OSU in a randomized assignment. Their personnel was trained to use Comfort Talk® to help patients who are claustrophobic, anxious, and/or cannot lie still to complete their tests at the onset of the study.
  Comfort Talk® Training: Personnel of MRI units will be trained in advanced rapport skills, patient-centered and hypnoidal language, correct use of suggestions and skills of tension diffusion. This will entail 16 hrs class room work, additional on-site post-training support, and access to a post-training support web module resulting in at least 20 hrs training.
- Control OSU: Three MRI sites at OSU were not trained in Comfort Talk®.
- Total: Total of all reporting groups
Arm/Group | Comfort Talk® Training OSU | Control OSU | Total
Number analyzed (Participants) | 0 | 0 | 0
Number analyzed (Imaging Slots) | 0 | 0 | 0
Age, Customized
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Equipment Utilization Q4FY15 = Baseline Quarter (OSU)
Description: Quarterly completion rate of MRIs as a proportion of scans completed per given number of imaging slots available
Time Frame: 1 quarter
Population: Imaging slots available in the quarter
Measure: Number; unit: Proportion of completed scans per slots
Units Other Than Participants: Imaging slots
Groups:
- Comfort Talk® Training: In the experimental group, MRI personnel is trained to use Comfort Talk® to help patients who are claustrophobic, anxious, and/or cannot lie still to complete their tests at the onset of the MRI scan.
  Comfort Talk® Training: Personnel of MRI units is trained in advanced rapport skills, patient-centered and hypnoidal language, correct use of suggestions and skills of tension diffusion. This will entail 16 hrs classroom work, additional on-site post-training support, and access to a post-training support web module resulting in at least 20 hrs training.
Arm/Group | Comfort Talk® Training | Control
Number analyzed (Participants) | 3940 | 3230
Number analyzed (Imaging slots) | 4754 | 4219
Proportion of completed scans per slots | 0.83 | 0.77

2. Primary Outcome: Equipment Utilization in Q1FY16 (OSU)
Description: Quarterly completion rate of MRIs as a proportion of scans completed per given number of imaging slots available
Time Frame: 1 quarter
Population: Participants completing their scans
Measure: Number; unit: Proportion of completed scans per slots
Units Other Than Participants: Imaging slots
Arm/Group | Comfort Talk® Training OSU | Control OSU
Number analyzed (Participants) | 3815 | 3032
Number analyzed (Imaging slots) | 4583 | 4144
Proportion of completed scans per slots | 0.832 | 0.732
Statistical Analysis 1: Comparison: Comfort Talk® Training OSU vs Control OSU; Comparison among trained and untrained sites; Test type: Superiority; p < 0.0001, Chi-squared, Corrected — Bonferroni-corrected p-values were used after multiplying the uncorrected p-value by 10
Statistical Analysis 2: Comparison: Comfort Talk® Training OSU; Change in the average quarterly completion rate as compared to the baseline quarter; Test type: Superiority; p = 0.3037, Chi-squared, Corrected — Bonferroni-corrected p-values were used after multiplying the uncorrected p-value by 10
Statistical Analysis 3: Comparison: Control OSU; Change in the average quarterly completion rate as compared to the baseline quarter; Test type: Superiority; p < 0.01, Chi-squared, Corrected — Bonferroni-corrected p-values were used after multiplying the uncorrected p-value by 10

3. Primary Outcome: Equipment Utilization in Q2FY16 (OSU)
Description: Quarterly completion rate of MRIs as a proportion of scans completed per given number of imaging slots available
Time Frame: 1 quarter
Population: Imaging slots available in the quarter
Measure: Number; unit: Proportion of completed scans per slots
Units Other Than Participants: Imaging Slots
Arm/Group | Comfort Talk® Training OSU | Control OSU
Number analyzed (Participants) | 3907 | 2857
Number analyzed (Imaging Slots) | 4659 | 4204
Proportion of completed scans per slots | 0.839 | 0.680
Statistical Analysis 1: Comparison: Comfort Talk® Training OSU vs Control OSU; Comparison among trained and untrained sites; Test type: Superiority; p < 0.0001, Chi-squared, Corrected — Bonferroni-corrected p-values were used after multiplying the uncorrected p-value by 10
Statistical Analysis 2: Comparison: Comfort Talk® Training OSU; Change in the average quarterly completion rate as compared to the baseline quarter; Test type: Superiority; p = 0.2010, Chi-squared — Bonferroni-correction was not done since the corrected p-value would be have been greater than 1
Statistical Analysis 3: Comparison: Control OSU; Change in the average quarterly completion rate as compared to the baseline quarter; Test type: Superiority; p < 0.001, Chi-squared — Bonferroni-corrected p-values were used after multiplying the uncorrected p-value by 10

4. Primary Outcome: Equipment Utilization in Q3FY16 (OSU)
Description: Quarterly completion rate of MRIs as a proportion of scans completed per given number of imaging slots available
Time Frame: 1 quarter
Population: Imaging slots available in the quarter
Measure: Number; unit: Proportion of completed scans per slots
Units Other Than Participants: Imaging slots
Arm/Group | Comfort Talk® Training OSU | Control OSU
Number analyzed (Participants) | 3928 | 2716
Number analyzed (Imaging slots) | 4647 | 4199
Proportion of completed scans per slots | 0.845 | 0.647
Statistical Analysis 1: Comparison: Comfort Talk® Training OSU vs Control OSU; Comparison among trained and untrained sites; Test type: Superiority; p < 0.0001, Chi-squared — Bonferroni-corrected p-values were used after multiplying the uncorrected p-value by 10
Statistical Analysis 2: Comparison: Comfort Talk® Training OSU vs Control OSU; Change in the quarterly equipment utilization rate as compared to the baseline quarter Q4FY15 over time and at sites; Test type: Superiority; p = 0.303, Chi-squared — Bonferroni-corrected p-values were used after multiplying the uncorrected p-value by 10. Chi-square analysis was used to assess equipment utilization at trained sites compared with untrained sites when stratifying by time (chi-square MH = 858.2)
Statistical Analysis 3: Comparison: Control OSU; Change in the average quarterly completion rate as compared to the baseline quarter; Test type: Superiority; p < 0.001, Chi-squared, Corrected — Bonferroni-corrected p-values were used after multiplying the uncorrected p-value by 10

5. Primary Outcome: Equipment Utilization Over All Quarters (OSU)
Description: Completion rates of MRIs as a proportion of scans completed per given number of imaging slots available
Time Frame: 4 quarters
Population: Imaging slots available
Measure: Number; unit: Proportion of completed scans per slots
Units Other Than Participants: Imaging slots
Arm/Group | Comfort Talk® Training OSU | Control OSU
Number analyzed (Participants) | 15590 | 11835
Number analyzed (Imaging slots) | 18643 | 16766
Proportion of completed scans per slots | 0.836 | 0.705
Statistical Analysis 1: Comparison: Comfort Talk® Training OSU vs Control OSU; Test type: Superiority; p < 0.0001, Chi-squared, Corrected — CMH test was used with time as a strata variable (rather than pooling all data together as in the regular chi-squared test). The CMH chi-squared value was 858.2, and the regular chi-squared value was 858.8; Bonferroni-corrected p-values were used after multiplying the uncorrected p-value by 10

6. Primary Outcome: Incompletions (Duke)
Description: Patients who cannot complete their scan
Time Frame: 9 months (3 months baseline, 6 months post training)
Population: Patients showing for their MRI scans
Measure: Count of Participants; unit: Participants
Groups:
- Baseline (Duke): Patients who show for their MRI scans prior to team Training in Comfort Talk®
- Post Comfort Talk® Training: Patient who show for their MRI scans after team training in Comfort Talk®
Arm/Group | Baseline (Duke) | Post Comfort Talk® Training
Number analyzed (Participants) | 4051 | 8879
Participants | 52 | 27
Statistical Analysis 1: Comparison: Baseline (Duke) vs Post Comfort Talk® Training; Test type: Superiority; p < 0.0001, Chi-squared

7. Secondary Outcome: No-shows in Q4FY15 = Baseline Quarter (OSU)
Description: Quarterly number of scheduled patients who do not show up for their appointments
Time Frame: 1 quarter
Population: Scheduled patients
Measure: Count of Participants; unit: Participants
Groups:
- Control: MRI sites are not be trained in Comfort Talk®.
  Please note that at OSU both trained and control sites had a baseline and three post-training periods.
  At Duke, the data in the initial baseline period became the control data in a pre to post comparison for reasons explained above. Therefore Duke has only 2 time period with the initial "Baseline" entered as "Control."
Arm/Group | Comfort Talk® Training | Control
Number analyzed (Participants) | 4158 | 3446
Participants | 218 | 216

8. Secondary Outcome: No-shows in Q1FY16 (OSU)
Description: Quarterly number of scheduled patients who do not show up for their appointments
Time Frame: 1 quarter
Population: Patients scheduled for MRI
Measure: Count of Participants; unit: Participants
Arm/Group | Comfort Talk® Training OSU | Control OSU
Number analyzed (Participants) | 4030 | 3246
Participants | 215 | 214
Statistical Analysis 1: Comparison: Comfort Talk® Training OSU vs Control OSU; Comparison among trained and untrained sites; Test type: Superiority; p = 0.2357, Chi-squared, Corrected — Bonferroni-corrected p-values were used after multiplying the uncorrected p-value by 10
Statistical Analysis 2: Comparison: Comfort Talk® Training OSU; Change in the quarterly no-shows as compared to the baseline quarter; Test type: Superiority; p = 0.8523, Chi-squared — No Bonferroni-correction
Statistical Analysis 3: Comparison: Control OSU; Change in the quarterly average no-show rate as compared to the baseline quarter at untrained sites; Test type: Superiority; p = 0.5883, Chi-squared — Bonferroni-correction was not done for this nonsignificant result since the corrected p-value would be have been greater than 1, which is not possible

9. Secondary Outcome: No-shows in Q2FY16 (OSU)
Description: Quarterly number of scheduled patients who do not show up for their appointments
Time Frame: 1 quarter
Population: Patients scheduled for MRI
Measure: Count of Participants; unit: Participants
Arm/Group | Comfort Talk® Training OSU | Control OSU
Number analyzed (Participants) | 4121 | 3070
Participants | 214 | 213
Statistical Analysis 1: Comparison: Comfort Talk® Training OSU vs Control OSU; Comparison among trained and untrained sites; Test type: Superiority; p = 0.0195, Chi-squared, Corrected — Bonferroni-corrected p-values were used after multiplying the uncorrected p-value by 10
Statistical Analysis 2: Comparison: Comfort Talk® Training OSU; Change in the quarterly no-shows compared to the baseline quarter; Test type: Superiority; p = 0.276, Chi-squared — No Bonferroni-correction
Statistical Analysis 3: Comparison: Control OSU; Change in the quarterly no-shows as compared to the baseline quarter at untrained sites; Test type: Superiority; p = 0.2764, Chi-squared — No Bonferroni-correction

10. Secondary Outcome: No-shows in Q3FY16 (OSU)
Description: Quarterly number of scheduled patients who do not show up for their appointments
Time Frame: 1 quarter
Population: Patients scheduled for MRI
Measure: Count of Participants; unit: Participants
Arm/Group | Comfort Talk® Training OSU | Control OSU
Number analyzed (Participants) | 4148 | 2931
Participants | 220 | 215
Statistical Analysis 1: Comparison: Comfort Talk® Training OSU vs Control OSU; Comparison among trained and untrained sites; Test type: Superiority; p < 0.01, Chi-squared, Corrected — Bonferroni-corrected p-values were used after multiplying the uncorrected p-value by 10
Statistical Analysis 2: Comparison: Comfort Talk® Training OSU; Change in the quarterly average no show rate as compared to the baseline quarter for trained sites; Test type: Superiority; p = 0.9012, Chi-squared — Bonferroni-correction was not done since the corrected p-value would be have been greater than 1
Statistical Analysis 3: Comparison: Control OSU; Change in the quarterly average no-show rate as compared to the baseline quarter for untrained sites; Test type: Superiority; p = 0.9065, Chi-squared, Corrected — Bonferroni-corrected p-values were used after multiplying the uncorrected p-value by 10

11. Secondary Outcome: Trend of No-shows Over All Quarters (OSU)
Description: Quarterly number of scheduled patients who do not show up for their appointments
Time Frame: 4 quarters
Population: Patients scheduled for MRI
Measure: Count of Participants; unit: Participants
Arm/Group | Comfort Talk® Training OSU | Control OSU
Number analyzed (Participants) | 16457 | 12693
Participants | 867 | 858
Statistical Analysis 1: Comparison: Comfort Talk® Training OSU vs Control OSU; Comparison among trained and untrained sites over time; Test type: Superiority; p < 0.0001, Chi-squared, Corrected — Bonferroni-corrected p-values were used after multiplying the uncorrected p-value by 10; CMH test with time as a strata variable was 28.7; chi-square value with pooling all data together was 28.6

12. Secondary Outcome: Patient Satisfaction Ranking in Q4FY15 = Baseline Quarter (OSU)
Description: Quarterly percentile rankings of patients' "Overall Assesment" of their satisfaction on a national clinical survey instrument (Press Ganey). Percentile rankings are benchmarked on 1,028 MRI sites nationally, given in raw scores between 0 (worst) to 100 (best). The percentile rankings are based on the number of participants returning surveys in each group.
Time Frame: 1 quarter
Population: Number of participants who returned surveys during that quarter.
Measure: Mean (Standard Deviation); unit: National Satisfaction Ranking
Arm/Group | Comfort Talk® Training OSU | Control OSU
Number analyzed (Participants) | 116 | 71
National Satisfaction Ranking | 42.3 (35.2) | 65.0 (36.7)

13. Secondary Outcome: Patient Satisfaction in Q1FY16 (OSU)
Description: as for outcome 12
Time Frame: 1 quarter
Population: Number of participants who returned surveys during that quarter.
Measure: Mean (Standard Deviation); unit: National Percentile Satisfaction Ranking
Arm/Group | Comfort Talk® Training OSU | Control OSU
Number analyzed (Participants) | 135 | 110
National Percentile Satisfaction Ranking | 71.0 (21.2) | 60.1 (41.7)

14. Secondary Outcome: Patient Satisfaction Ranking in Q2FY16 (OSU)
Description: as for outcome 12
Time Frame: 1 quarter
Population: Number of participants who returned surveys during that quarter.
Measure: Mean (Standard Deviation); unit: National Percentile Satisfaction Ranking
Arm/Group | Comfort Talk® Training OSU | Control OSU
Number analyzed (Participants) | 138 | 106
National Percentile Satisfaction Ranking | 75.3 (16.8) | 42.3 (40.1)

15. Secondary Outcome: Patient Satisfaction Ranking in Q3FY16 (OSU)
Description: as for outcome 12
Time Frame: 1 quarter
Population: Number of participants who returned surveys during that quarter.
Measure: Mean (Standard Deviation); unit: National Percentile Satisfaction Ranking
Arm/Group | Comfort Talk® Training OSU | Control OSU
Number analyzed (Participants) | 158 | 87
National Percentile Satisfaction Ranking | 76.7 (16.9) | 36 (41.7)

16. Secondary Outcome: Oral Sedation Rate (Duke)
Description: Patients who receive medical sedation on site
Time Frame: 9 months (3 months baseline, 6 months post training)
Population: Patients showing for their MRI scans
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline (Duke) | Post Comfort Talk® Training
Number analyzed (Participants) | 4051 | 8879
Participants | 100 | 128
Statistical Analysis 1: Comparison: Baseline (Duke) vs Post Comfort Talk® Training; Test type: Superiority; p < 0.0001, Chi-squared

17. Secondary Outcome: IV Sedation Rate (Duke)
Description: Number of patients who receive intravenous (IV) sedation on site
Time Frame: 9 months (3 months baseline, 6 months post training)
Population: Patients showing for their MRI scans
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline (Duke) | Post Comfort Talk® Training
Number analyzed (Participants) | 4051 | 8879
Participants | 103 | 196
Statistical Analysis 1: Comparison: Baseline (Duke) vs Post Comfort Talk® Training; Test type: Superiority; p = 0.2396, Chi-squared

18. Secondary Outcome: General Anesthesia Rate (Duke)
Description: Number of patients who receive general anesthesia on site
Time Frame: 9 months (3 months baseline, 6 months post training)
Population: Patients showing for their MRI scans
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline (Duke) | Post Comfort Talk® Training
Number analyzed (Participants) | 4051 | 8879
Participants | 29 | 55
Statistical Analysis 1: Comparison: Baseline (Duke) vs Post Comfort Talk® Training; Test type: Superiority; p = 0.5267, Chi-squared

19. Secondary Outcome: Disruptive Motion (Duke)
Description: Patients on site who disrupt the scan by motion
Time Frame: 9 months (3 months baseline, 6 months post training)
Population: Patients showing for their MRI scans
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline (Duke) | Post Comfort Talk® Training
Number analyzed (Participants) | 4051 | 8879
Participants | 42 | 11
Statistical Analysis 1: Comparison: Baseline (Duke) vs Post Comfort Talk® Training; Test type: Superiority; p < 0.0001, Chi-squared

20. Secondary Outcome: No-shows (Duke)
Description: Scheduled patients who do not show for their MRI examinations.
Time Frame: 9 months (3 months baseline, 6 months post training)
Population: Patients scheduled for MRI scans
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline (Duke) | Post Comfort Talk® Training
Number analyzed (Participants) | 4446 | 9658
Participants | 395 | 779
Statistical Analysis 1: Comparison: Baseline (Duke) vs Post Comfort Talk® Training; Test type: Superiority; p < 0.0001, Chi-squared

ADVERSE EVENTS:
Time Frame: One year starting with the training
Description: Adverse events were monitored during the training days of the MRI teams. Then assessment was non-systematic in that we would have reported adverse events if they had become known or being collected after training. Patients at risk were only those in the post-training period who showed up at the facility including those who completed their scans and also those who did not.
  Number of deaths was not specifically monitored.
Groups:
- Comfort Talk® Training (OSU): Three MRI clinical sites form the experimental group. Their personnel was trained to use Comfort Talk® to help patients who are claustrophobic, anxious, and/or cannot lie still to complete their tests at the onset of the study.
  Comfort Talk® Training: Personnel of MRI units will be trained in advanced rapport skills, patient-centered and hypnoidal language, correct use of suggestions and skills of tension diffusion. This will entail 16 hrs classroom work, additional on-site post-training support, and access to a post-training support web module resulting in at least 20 hrs training.
- Control (OSU): Three MRI sites were not trained in Comfort Talk®.
- Baseline = Control (Duke): Data from 6 Duke sites at baseline were used as the control in a pre- to post-training comparison
- Comfort Talk® Training (Duke): The same 6 Duke sites represented at baseline formed the experimental group after Comfort Talk training in a pre- to post- training comparison
Arm/Group | Comfort Talk® Training (OSU) | Control (OSU) | Baseline = Control (Duke) | Comfort Talk® Training (Duke)
All-Cause Mortality (participants affected / at risk) | 0/11650 | 0/8605 | 0/4446 | 0/9658
Serious Adverse Events (participants affected / at risk) | 0/11650 | 0/8605 | 0/4446 | 0/9658
Other Adverse Events (participants affected / at risk) | 0/11650 | 0/8605 | 0/4446 | 0/9658

LIMITATIONS AND CAVEATS:
Because of considerable staff cuts at Duke right personnel rotated among all sites so that randomization based on training could not be maintained. Therefore a pre/post training comparison was done. OSU collected data electronically, Duke by diary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2015-08-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT02427737/Prot_000.pdf